CLINICAL TRIAL: NCT06233799
Title: Randomized, Placebo-Controlled, Multi-Site Trial of Extended-Release Naltrexone Injection/Bupropion XL Tablets in the Treatment of Methamphetamine Use Disorder
Brief Title: Trial of Naltrexone/Bupropion for the Treatment of Methamphetamine Use Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA/VA CS #1036
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Methamphetamine-dependence; Methamphetamine Abuse
MeSH Terms: interventions — vivitrol; Tablets; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- XR-NTX/BUP-XL (Experimental): Participants randomized to the (XR-NTX/BUP-XL) arm will receive 450 mg of once-daily oral extended-release bupropion tablets and once every three weeks (Weeks 1, 4, 7, and 10) injections of extended-release naltrexone (Vivitrol®)
  Interventions: Drug: extended-release naltrexone (XR-NTX); Drug: extended release bupropion (BUP-XL) tablets (BUP-XL)
- PLB/PLB (Placebo Comparator): Participants randomized to the PLB arm will receive once-daily placebo tablets and once every three weeks (Weeks 1, 4, 7, and 10) placebo injections.
  Interventions: Drug: iPLB; Drug: oPLB

INTERVENTIONS:
Drug: extended-release naltrexone (XR-NTX) — Once per three weeks injections of extended-release naltrexone
  Other Names: Vivitrol
  Arms: XR-NTX/BUP-XL
Drug: extended release bupropion (BUP-XL) tablets (BUP-XL) — Daily oral extended release bupropion tablets
  Other Names: Wellbutrin
  Arms: XR-NTX/BUP-XL
Drug: iPLB — Once per three weeks injections of placebo
  Other Names: Placebo injections
  Arms: PLB/PLB
Drug: oPLB — Daily oral placebo tablets
  Other Names: Placebo tablets
  Arms: PLB/PLB

SUMMARY:
The primary objective of this study is to evaluate the efficacy of extended release naltrexone plus bupropion XL (XR-NTX/BUP-XL) compared to matched injectable and oral placebo (iPLB/oPLB) in reducing methamphetamine (MA) use in individuals with moderate or severe methamphetamine use disorder (MUD) seeking to stop or reduce MA use.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized clinical trial in which 360 individuals with moderate or severe MUD will be randomly assigned at a 1:1 ratio to receive either 1) extended release naltrexone (XR-NTX; as Vivitrol®) plus once daily oral extended release bupropion (BUP-XL) tablets (the XR-NTX/BUP-XL group) or 2) both the matching injection placebo (iPLB) and once daily oral placebo (oPLB) tablets (the iPLB/oPLB group). The study intervention consists of a 12-week treatment phase. It is hypothesized that the XR-NTX/BUP-XL arm will be associated with a greater number of "responders," defined as participants who provide at least 3 MA-negative urine drug screens (UDS) out of 4 samples obtained during the evaluation period (i.e., Weeks 11-12) of the 12-week long treatment phase, relative to the iPLB/oPLB arm. Secondary objectives include evaluating the effect of the extended release naltrexone plus bupropion XL (XR-NTX/BUP-XL) arm compared to the iPLB/oPLB arm on safety, other substance use outcomes, depression scores, quality of life, overall functioning, clinic attendance, and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 to 65 years of age;
2. Meets DSM-5 criteria for moderate or severe MUD (4 or more criteria);
3. Is interested in reducing or stopping MA use;
4. Is able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study;
5. Self-reports MA use on 18 or more days in the 30-day period prior to consent using the Timeline Followback (TLFB);
6. Provides at least 2 urine samples positive for MA out of up to 3 tests, which will occur at least 2 days apart within a 10-day period;
7. If assigned as female at birth and/or currently has a uterus, is not pregnant, agrees to use acceptable birth control methods, and have periodic urine pregnancy testing done during participation in the study unless documentation of hysterectomy provided;
8. Is not physically dependent on opioids and meets subjective and objective measures of being opioid-free prior to naltrexone injection per study medical clinician's determination, including, if clinically required, a negative naloxone challenge;
9. Is willing to comply with all study procedures and medication instructions;
10. Agrees to use a smartphone app (downloaded for free to own device or on a study provided smartphone device) to take daily videos of medication dosing.

Exclusion Criteria:

1. Has an acute medical or psychiatric disorder that would, in the judgment of the study medical clinician, make participation difficult or unsafe;
2. Has suicidal or homicidal ideation that requires immediate attention;
3. Has a history of epilepsy, seizure disorder, or head trauma with neurological sequelae (e.g., loss of consciousness that required hospitalization); current anorexia nervosa or bulimia; or any other conditions that increase seizure risk in the opinion of the study medical clinician;
4. Has evidence of second or third degree heart block, atrial fibrillation, atrial flutter, prolongation of the QTc, or any other finding on the screening ECG that, in the opinion of the study medical clinician, would preclude safe participation in the study;
5. Has Stage 2 hypertension as determined by the study medical clinician (e.g., greater than or equal to 160/100 in 2 out of 3 readings during screening);
6. Has any elevated bilirubin test value per laboratory criteria OR any other liver function test (LFT) value > 5 times the upper limit of normal per laboratory criteria;
7. Has a platelet count <100 x 10exp3/microliter;
8. Has a body habitus that precludes gluteal intramuscular injection of XR-NTX in accordance with the administration equipment (needle) and procedures;
9. Has a known allergy or sensitivity to bupropion, naloxone, naltrexone, PLG (polyactideco-glycolide), carboxymethylcellulose or any other component of the XR-NTX diluents;
10. Has been in a prior study of pharmacological or behavioral treatment for MUD within 6 months of study consent;
11. Has taken an investigational drug in another study within 30 days of study consent;
12. Has been prescribed and taken naltrexone or bupropion within 30 days of study consent;
13. Is concurrently enrolled in formal behavioral or pharmacological Substance Use Disorder (SUD) treatment services;
14. Is receiving ongoing treatment with tricyclic antidepressants, xanthines (i.e., theophylline and aminophylline), systemic corticosteroids, nelfinavir, efavirenz, chlorpromazine, MAOIs, central nervous system stimulants (e.g., Adderall, Ritalin, etc.), or any medication that, in the judgment of the study medical clinician, could interact adversely with study medications;
15. Has a current pattern of alcohol, benzodiazepine, or other sedative hypnotic use which would preclude safe participation in the study as determined by the study medical clinician;
16. Requires treatment with opioid-containing medications (e.g., opioid analgesics) during the study period;
17. Has a surgery planned or scheduled during the study period;
18. Is currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or other situation (e.g., unstable living arrangements) that could prevent participation in the study or in any study activities;
19. If assigned as female at birth and/or currently has a uterus, is currently pregnant, breastfeeding, or planning on conception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with at least 75% methamphetamine-negative urine drug screen tests during the evaluation period (i. e., Weeks 11-12) | 2 weeks (i. e., Weeks 11-12)
  Participants will be administered four urine drug screen tests (two tests/week) during the evaluation period. (i.e., Weeks 11-12).

SECONDARY OUTCOMES:
safety measured as frequency and severity of adverse events (AEs) | 16 weeks (12 week treatment plus followup)
  adverse events (AEs), clinical lab tests, suicidality
Severity of Craving as measured by Visual Analog Scale | 16 weeks (12 week treatment plus followup)
  Craving score as assessed by Visual Analog Scale that ranges from 0 (no craving) to 100 (most intense craving possible). The Visual Analog Scale will be completed at each screening visit, twice weekly throughout the treatment phase, and at the Week 14 and 16 follow-up visits.
Severity of Depression as assessed by the Patient Health Questionnaire-9 | 16 weeks (12 week treatment plus followup)
  Diagnostic criteria for major depression, severity and frequency of depressive symptoms, presence of suicidal ideation, and functional impairment related to depression will be assessed by the Patient Health Questionnaire-9 (Kroenke et al., 2001)
Treatment Effectiveness as measured by the Treatment Effectiveness Assessment | 16 weeks (12 week treatment plus followup)
  The Treatment Effectiveness Assessment (TEA; Ling et al., 2012) is a 4-item self-administered assessment to document changes in four life domains: substance use, personal responsibilities, health, and community. The TEA will be collected at screening, mid-treatment (Week 6 visit 2), end-of-treatment (Week 12 visit 2), and follow-up (Weeks 14 and 16).
Quality of Life as measured by PROMIS® Profile 29 for adults | 16 weeks (12 week treatment plus followup)
  The instrument includes 29 self-administered questions from the PROMIS® Profile 29 for adults. The quality of life questions include physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain intensity over the past 30 days. Each question, except for the pain intensity question, is measured on a 5-point scale. Quality of Life will be assessed at screening, mid-treatment (Week 6 visit 2), end-of-treatment (Week 12 visit 2), and follow-up (Weeks 14 and 16).

CONTACTS AND LOCATIONS:
Overall Officials: Raul Mandler, MD, Principal Investigator — NIDA/NIH
Locations (11):
- United States (11):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - CODA, Portland, Oregon
  - MUSC/BHS, Pickens, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
Investigators don't plan to make individual participant data (IPD) available to other researchers.